CLINICAL TRIAL: NCT04394676
Title: The Impact of Low Pressure Pneumoperitoneum in Robotic Assisted Radical Prostatectomy: A Prospective Randomized Controlled Trial II
Brief Title: The Impact of Low Pressure Pneumo in RARP II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Metro Health, Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB2020-007
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Radical Prostatectomy; Robotic Assisted Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduction in Pressure (Experimental): This group receives 12mm Hg of pneumoperitoneum pressure during robotic assisted radical prostatectomy.
  Interventions: Procedure: Pressure applied during RARP
- Standard Amount of Pressure (Active Comparator): This group receives 15mm Hg of pneumoperitoneum pressure during robotic assisted radical prostatectomy (RARP). This pressure is the standard amount used for all RARP procedures.
  Interventions: Procedure: Pressure applied during RARP

INTERVENTIONS:
Procedure: Pressure applied during RARP — Patients will be randomly assigned to undergo RARP either at a pneumoperitoneum pressure of 12 mmHg (experimental) or 15mm Hg (standard technique).

SUMMARY:
The purpose of this study is to evaluate clinical significance of low pressure pneumoperitoneum during robotically assisted radical prostatectomy (RARP).

DETAILED DESCRIPTION:
Laparoscopic and robotic surgery has revolutionized post-operative outcomes across surgical specialties. However, the use of pneumoperitoneum comes with known risks given the change in physiological parameters that accompany its utilization. The effects of increased intra-abdominal pressure on cardiopulmonary function has been well documented. Increased pressure on the large vessels may lead to decreased cardiac output and thereby decreased blood flow to various organ systems and cause irreversible damage. Some studies have advocated lower pressures to further optimize cardiopulmonary parameters. McDougall, et. al, for instance, demonstrated a significant reduction in oliguria when pressures of 10mm Hg were used. The purpose of this study is to evaluate the effect of using lower pressure pneumoperitoneum in the abdominal cavity during RARP. The investigators hypothesize that low pressure pneumoperitoneum has a multitude of clinical benefits due to improved physiologic parameters including a reduction in the occurrence of post-operative ileus, reduced need for narcotics post operatively, and a decrease in cardiopulmonary complications. A previously completed study concluded a reduction in post-operative ileus at a pneumoperitoneum pressure of 8 mm Hg vs 12 mm Hg. This new study will evaluate the standard pneumoperitoneum pressure of 15 mm Hg vs 12 mm Hg in order to validate the previous study vs the standard pneumoperitoneum pressure.

The study is a prospective randomized blinded cohort study. Patients who meet eligibility criteria will be randomly assigned to undergo RARP at a pneumoperitoneum pressure of 15mm Hg or 12mm Hg. This will be done by computer generated randomization protocol. Surgeon and patients will be blinded to the pneumoperitoneum pressure used. A cover will be placed over the insufflation system so that the surgeon(s) are not able to visualize the pneumoperitoneum used during the procedure. The remainder of the procedure will be carried out based on current standard of care. All patients will be admitted post operatively and the same standardized orderset in EPIC EHR will be used for all patients in order to control for other factors, such as opioid use, to control for confounders.

ELIGIBILITY:
Inclusion Criteria:

- Male 40 years of age or older

* Diagnosis of prostate cancer
* Have been evaluated to be fit for proposed surgery
* Patients able to consent

Exclusion Criteria:

- Patients unable to consent (cognitively impaired)

• Non-English speaking

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of Post-Operative Ileus | An average of 3 days
  Reduction in the occurrence of Post-Operative Ileus after RARP

SECONDARY OUTCOMES:
Reduction in narcotic use | An average of 3 days
  Reduction in the need for narcotics post operatively
Reduction in Estimated Blood Loss during RARP | An average of 1 hour
  Reduced blood loss during robot assisted radical prostatectomy
Reduction in post operative complications as measured by Clavien-Dindo Complication Score | Up to 30 days after procedure
  Reduction in post operative complications as measured by Clavien-Dindo Complication Score

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maatman, DO, Principal Investigator — Michigan Urological Clinic
Locations (1):
- Metro Health-University of Michigan Health, Wyoming, Michigan, United States

IPD SHARING:
Plan to Share IPD: No